CLINICAL TRIAL: NCT06398600
Title: Analgesic Effect of Ultrasound Guided Caudal Block Versus Quadratus Lumborum Plane Block in Lumbar Spine Surgery in Adult Patients: A Double Blinded Prospective Comparative Study
Brief Title: Caudal Block Versus Quadratus Lumborum Plane Block in Lumbar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed mahmoud, Associate professor of anesthesia, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M 696
Record Dates: First submitted 2024-04-26; First posted 2024-05-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Spondylolisthesis; Facet Joint Hypertrophy; Spinal Canal Stenosis
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be achieved using computer-generated random numbering of each study patient. opaque sealed envelopes will be used and opened in the operating room by a anesthesia resident who will be blinded to the study. The patient and researcher who collects the data after the block will be blinded to the study group. All study outcomes will be evaluated by a dedicated anesthesiologist who will be blinded to the group allocation. Patients will be randomized into three groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caudal block group (Active Comparator): This group of patient receiving caudal block in prone position before the operation.
  Interventions: Procedure: Caudal
- Quadratus lumborum plane block (Active Comparator): This group of patient receiving quadratus lumborum plane block in prone position before the operation.
  Interventions: Procedure: Quadratus lumborum plane block
- controlled group (No Intervention): this group of patient will not receive any blocks, only undergoing operation under general anesthesia and receive only 1 g paracetamol 30 min before end of operation

INTERVENTIONS:
Procedure: Caudal — In the prone position , linear transducer will be first positioned transversely on the middle line. The two sacral cornua appear as two hyperechoic structures ,two hyperechoic band structures are present between the two sacral cornua. The superficial is the sacrococcygeal ligament (SCL) and the deep is the dorsal surface of the sacrum. The sacral hiatus is a hypoechoic area between two band-like hyperechoic structures. In longitudinal view, the block needle will be inserted using the in plane technique .The block needle can be visualized in real time piercing the SCL entering the hiatus but cannot be visualized beyond the apex of the hiatus. It is therefore proposed to limit the extension of the needle tip beyond the tip of the sacral hiatus to 5 mm to avoid perforating the dura mater. After the needle is inserted in the caudal canal, 20 ml of 0.25% bupivacaine will be injected.
  Arms: Caudal block group
Procedure: Quadratus lumborum plane block — The patient is placed in the prone position , under aseptic conditions with the sterile convex probe is placed in a transverse view at the triangle of the QL muscle and the middle thoracolumbar fascia. The projected needle path is advanced in-plane until the needle tip is visualized between the middle thoracolumbar fascia and the QL muscle . After confirming the location of the needle with 2-3 ml of saline and then aspiration, 20 ml of 0.25% bupivacaine is injected in this plane with confirmation by visualizing hydro dissection . the procedure is applied to the opposite side using the same dose to achieve bilateral block.
  Arms: Quadratus lumborum plane block

SUMMARY:
Postoperative pain is a common complication after lumbar spine surgery due to inherent tissue damage during surgical procedures.

Many analgesic options have been explored. Opioid analgesics carry the risk of respiratory depression.

Nonsteroidal anti-inflammatory drugs (NSAIDs) are popular and widely used as first-line treatment for acute pain following spinal surgery, but can provide inadequate analgesia. High doses of NSAIDs have also been linked to non-unions in spinal fusion surgery.

Patient-controlled analgesia or epidural injection analgesia are usually used. One of US guided regional anesthesia methods is the ultrasound-guided caudal block that was first described by Klocke and colleagues in 2003.

One of the more recent techniques that has been described recently is quadratus lumborum plane block(QLB),that is posterior abdominal wall fascial plane block first described by Blanco in 2007.In this study we will compare between analgesic effect of ultrasound guided caudal block to that of ultrasound guided quadratus lumborum plane block as well as safety of both modalities in adult patients undergoing lumbar spine fixation surgeries.

DETAILED DESCRIPTION:
This study will be conducted at Fayoum University Hospital after the approval of the local institutional ethics committee and local institutional review board. The study design will be a randomized, double-blind, controlled study. A detailed informed consent form will be signed by eligible patients prior to enrollment and randomization.

Inclusion criteria:

Anesthesia procedure Patients will be randomly allocated into one of three parallel groups (37 in each group) based on sample size. Randomization will be achieved using computer-generated random numbering of each study patient. opaque sealed envelopes will be used and opened in the operating room by a anesthesia resident who will be blinded to the study. The patient and researcher who collects the data after the block will be blinded to the study group. All study outcomes will be evaluated by a dedicated anesthesiologist who will be blinded to the group allocation. Patients will be randomized into three groups.

Group (D) patients who will receive caudal block. Group (QL) patients who will receive posterior quadratus lumborum plane block. Group (C) patients who will not receive any blocks. Preoperative assessment A preoperative patient visit will be done for medical history taking, clinical examination, reassurance, and explaining the method of anesthesia. The study protocol, caudal block, quadratus lumborum plane block and the numerical pain rating score score will be explained to each patient during the preanesthetic counselling. The patient's back will be examined to detect any spinal deformities . Patients will fast for about 6 to 8 hours for solid meals , for 4 hours for non clear liquids and for 2 hours for clear liquids before surgery.

Intraoperative management Monitoring equipment will be connected to the patients included pulse oximetry, non-invasive blood pressure monitoring, five-lead electrocardiogram and capnography. IV access will be established. Patients in the three groups will receive general anesthesia after 5 minutes of pre oxygenation with 100% O2. Anesthesia will be induced with intravenous fentanyl 1mcg/kg, propofol 2 mg/kg and atracurium 0.5 mg/kg. After oral endotracheal intubation, anesthesia will be maintained with isoflurane (1.2%_1.5%) in oxygen _air mixture and atracurium 0.1mg/kg with interval about 20 min.

Block technique After stabilizing the patient hemodynamics, caudal block or quadratus lumborum plane block will be performed in the prone position prior to the skin incision after aseptic preparation of injection area.

Petit between the iliac crest and the costal margin where the trans abdominal muscle is identified . The transducer is then slid posterior until the trans abdominal muscle posterior aponeurosis is identified adjacent to Caudal block

The patient is placed in the prone position typically, a linear transducer is sufficient for the most caudal epidural injection; However, obese patients may require curved transducer. The Ultrasound transducer of (LOGIQ P7 ultrasound) will be first positioned transversely on the midline to obtain a transverse view of the sacral hiatus. The two sacral cornua appear as two hyperechoic structures ,two hyperechoic band structures are present between the two sacral cornua. The superficial is the sacrococcygeal ligament (SCL) and the deep is the dorsal surface of the sacrum. The sacral hiatus is a hypoechoic area between two band-like hyperechoic structures. At this level, the ultrasound probe is rotated 90 degrees to obtain a longitudinal view of the sacral hiatus. in the longitudinal view, the block needle will be inserted using the in plane technique .The block needle can be visualized in real time piercing the SCL entering the hiatus but cannot be visualized beyond the apex of the hiatus. It is therefore proposed to limit the extension of the needle tip beyond the tip of the sacral hiatus to 5 mm to avoid perforating the dura mater, since the distance between the tip of the sacral hiatus and the tip of the dural sac can be less than 6 mm .After the needle is inserted in the caudal canal, 20 ml of 0.25% bupivacaine will be injected. Presence of unidirectional flow, defined as dominant color on color Doppler image, In longitudinal view of sacral hiatus during injection will be reported to be predictive of successful caudal injection and comparable treatment outcomes.

Quadratus Lumborum Plane Block The patient is placed in the prone position , under aseptic conditions with the sterile convex probe is placed in a transverse view at the triangle of the QL muscle and the middle thoracolumbar fascia. The projected needle path is advanced in-plane until the needle tip is visualized between the middle thoracolumbar fascia and the QL muscle .After confirming the location of the needle with 2-3 ml of saline and then aspiration, 20 ml of 0.25% bupivacaine is injected in this plane with confirmation by visualizing hydro dissection . the procedure is applied to the opposite side using the same dose to achieve bilateral block.

Maintenance and recovery Inadequate analgesia that is predicted by increase of heart rate or mean arterial blood pressure by more than 20% of baseline will be managed by 0.5mcg/Kg of fentanyl. Total IV consumption of fentanyl will be recorded. All patients will receive 4mg ondansetron and 1 g paracetamol intravenously 30 minutes before the end of the operation. At the end of surgery, all patients will undergo reversal of muscle relaxation with neostigmine 0.05 mg/kg and atropine 0.01 mg/kg.

After recovery from anesthesia, patients will be transferred to recovery room where heart rate, respiratory rate, saturation and systolic, diastolic and mean arterial blood pressure will be monitored. Quality of analgesia will be assessed using numerical pain rating scale (NPRS) Assessment will be performed at admission to the recovery room, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 18 h, and 24 h postoperative. Rescue analgesia in the form of pethidine 0.5 mg/kg will be administered if is pain moderate to severe according to NPRS≥4 . Time to the 1st rescue analgesic request is recorded.

Also intraoperative or postoperative complications will be recorded such as local anesthetic toxicity, hypotension, nausea, vomiting as well as neurologic complications such as weakness, numbness or any neurological deficits. Also operative time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-60 years old), of either gender undergoing elective lumbar spine fixation surgery.
2. Patients with American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

1. Include patients who refuse.
2. Patients with contraindications to regional anesthesia (eg, local infection at site of injection, coagulation abnormalities).
3. Patients with spinal deformities or previous lumbar disc surgeries.
4. Allergy to local anesthetics, mental disorders as well as drug abuse.
5. BMI more than 35

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesic request. | first 24 hours
  duration between time of introducing intervention and time of first analgesic request

SECONDARY OUTCOMES:
The postoperative numerical pain rating score for 24 h | for first 24 hours
  The numerical pain rating score is an 11-point scale scored from 0_10 where (0) equal no pain, (1_3) equal mild pain,( 4_6) equal moderate pain and (7_10) equal severe pain.
Total opioid consumption used in first 24 hours . | for first 24 hours
  total dose of opioids consumed
Intraoperative fentanyl consumption. | during intra operative period
  dose of fentanyl consumed
Intraoperative heart rate every 15 minutes. | during intra operative period
  Heart rate is measured every 15 minutes during the whole duration of operation
Intraoperative blood pressure every 15 minutes | during intra operative period
  Blood pressure is measured every 15 min during the whole duration of operation
postoperative heart rate every 2h for 24h. | for first 24 hours
  Heart rate is measured every 2 hours after the end of operation
postoperative blood pressure every 2h for 24h. | for first 24 hours
  Blood pressure is measured every 2 hours after the end of operation
Complications related as local anesthetic toxicity, nausea and vomiting. | for first 24 hours
  any complications detected

CONTACTS AND LOCATIONS:
Overall Officials: Atef Mohamed, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klocke R, Jenkinson T, Glew D. Sonographically guided caudal epidural steroid injections. J Ultrasound Med. 2003 Nov;22(11):1229-32. doi: 10.7863/jum.2003.22.11.1229. PMID 14620894
- [Background] Korgvee A, Junttila E, Koskinen H, Huhtala H, Kalliomaki ML. Ultrasound-guided quadratus lumborum block for postoperative analgesia: A systematic review and meta-analysis. Eur J Anaesthesiol. 2021 Feb 1;38(2):115-129. doi: 10.1097/EJA.0000000000001368. PMID 33186305
- [Background] Chen CP, Tang SF, Hsu TC, Tsai WC, Liu HP, Chen MJ, Date E, Lew HL. Ultrasound guidance in caudal epidural needle placement. Anesthesiology. 2004 Jul;101(1):181-4. doi: 10.1097/00000542-200407000-00028. PMID 15220789
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561